CLINICAL TRIAL: NCT00001226
Title: Lipoprotein Metabolism in Normal Volunteers and Dyslipoproteinemic Patients (Stable Isotopes)
Brief Title: Lipoprotein Metabolism in Normal Volunteers and Patients With Abnormal Levels of Lipoproteins
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 870207; 87-H-0207
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-03

CONDITIONS: Healthy; Hyperlipoproteinemia
Keywords: Nonradioactive Isotopes; Lipoprotein Kinetics; Apolipoproteins; Dyslipoproteinemia; Healthy Volunteers
MeSH Terms: conditions — Hyperlipoproteinemias; Dyslipidemias

SUMMARY:
Researchers plan to study the fat-rich particles, called lipoproteins, which circulate in the blood. This study is designed to improve understanding of normal, as well as abnormal, lipoprotein metabolism and the role it plays in the development of hardening of the arteries (atherosclerosis).

Patients participating in this study will receive an intravenous (directly into the vein) injection of a small amount of specially prepared amino acids. The amino acids being injected are the same amino acids present in a normal diet. The amount of amino acid given will be less than the amount eaten in a protein-rich meal. The amino acids will be labeled with nonradioactive heavy isotopes which are also present in the environment n low amounts.

Patients participating in the study will be required to have blood samples taken, and provide urine samples throughout the course of the study. In addition, patient will be required to follow a specially formulated diet. Patients will be weighed throughout the course of the study.

DETAILED DESCRIPTION:
Apolipoproteins regulate the metabolism of lipids and lipoproteins in plasma of humans. In order to investigate the roles of apolipoproteins in these processes, we plan to quantitate the kinetics of the metabolism of apolipoproteins utilizing nonradioactive isotope labeled amino-acids.

ELIGIBILITY:
The subjects for these investigations will be either healthy normal volunteer control subjects or patients who have a dyslipoproteinemia.

Subjects must be 18-80 years old.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 1987-12; Study Completion 2002-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Gordon T, Castelli WP, Hjortland MC, Kannel WB, Dawber TR. High density lipoprotein as a protective factor against coronary heart disease. The Framingham Study. Am J Med. 1977 May;62(5):707-14. doi: 10.1016/0002-9343(77)90874-9. PMID 193398
- [Background] Blankenhorn DH, Nessim SA, Johnson RL, Sanmarco ME, Azen SP, Cashin-Hemphill L. Beneficial effects of combined colestipol-niacin therapy on coronary atherosclerosis and coronary venous bypass grafts. JAMA. 1987 Jun 19;257(23):3233-40. PMID 3295315
- [Background] Brown MS, Goldstein JL. A receptor-mediated pathway for cholesterol homeostasis. Science. 1986 Apr 4;232(4746):34-47. doi: 10.1126/science.3513311. No abstract available.